CLINICAL TRIAL: NCT04891575
Title: Heart of the Family: A Cardiovascular Disease and Type 2 Diabetes Risk Reduction Intervention in High-Risk Rural Families
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gia Mudd (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor-Investigator, Gia Mudd, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 60980; 1R01NR019456-01 (NIH)
Record Dates: First submitted 2021-05-13; First posted 2021-05-18 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus, Type 2; Cardiovascular Diseases
Keywords: lifestyle modification; rural; Hispanic; non-Hispanic; dyad; family; risk reduction
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, intervention providers and assessors are blinded to which arm is the active intervention and which is the active comparator and are blinded to hypotheses regarding group differences.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Control Arm (Active Comparator): An index participant with 2 or more risk factors for cardiovascular disease or type 2 diabetes who is randomized to this arm will attend 8 weekly educational sessions focused on self-management of risk factors and engagement in healthy behaviors for risk reduction. The index participant will attend the sessions as an individual and will receive standard individual-focused lifestyle modification education.
  Interventions: Behavioral: Active Control Intervention educational sessions
- Family Dyad Arm (Experimental): An index participant with 2 or more risk factors for cardiovascular disease or type 2 diabetes and a co-participating family member will together attend 8 weekly educational sessions focused on self-management of risk factors and engagement in healthy behaviors for risk reduction. The dyadic intervention sessions also incorporate family-focused throughout each session to encourage dyadic support.
  Interventions: Behavioral: Family Dyad Intervention

INTERVENTIONS:
Behavioral: Active Control Intervention educational sessions — The participant will attend 8 sessions that provide type 2 diabetes (T2D) and cardiovascular (CVD) risk reduction and lifestyle modification education focused on CVD and T2D risk factor reduction through promotion of participant self-management. Education will concentrate on healthy eating, physical activity, stress reduction, and other lifestyle risk reduction recommendations.
  Arms: Active Control Arm
Behavioral: Family Dyad Intervention — The participant and a co-participating family member will attend 8 sessions that provide type 2 diabetes (T2D) and cardiovascular (CVD) risk reduction and lifestyle modification education focused on CVD and T2D risk factor reduction through promotion of participant self-management. Education will concentrate on healthy eating, physical activity, stress reduction, and other lifestyle risk reduction recommendations.
  Arms: Family Dyad Arm

SUMMARY:
Rural populations in the U.S. are disproportionately burdened by cardiovascular disease and type 2 diabetes. Lifestyle modification interventions are needed that support long-term engagement in risk-reducing health behaviors. This trial will study the effects of a family-focused, lifestyle intervention that is culturally tailored for use with rural Hispanic and non-Hispanic adults. If successful, this community-based intervention has significant potential for broad dissemination to reduce cardiovascular disease and type 2 diabetes health disparities in rural U.S. communities.

DETAILED DESCRIPTION:
The Heart of the Family study is a randomized controlled trial conducted to examine if a virtual lifestyle modification intervention is more effective in reducing risk for type 2 diabetes (T2D) and cardiovascular disease (CVD) when it is delivered to family dyads or to individuals and to compare intervention effects in Hispanic and non-Hispanic rural-dwelling adults at-risk for T2D or CVD. The Heart of the Family study will enroll 360 participants - 180 Hispanics and 180 non-Hispanics - from rural communities who have two or more risk factors for T2D or CVD. Participants will be randomized to participate as an individual or with a family member who may or may not be at risk for T2D or CVD or may or may not have diagnosed T2D or CVD for a total of 540 participants. The interventions for both groups will be provided by community health workers using a virtual platform. Both groups will receive eight educational sessions about healthy lifestyle behaviors and support to address personal and environmental barriers to engaging in healthy behaviors. After the eight sessions, the community health workers will follow up with participants once a month by phone over the next 12 months. Primary outcomes include short-term and long-term impact of the family-focused active intervention compared to the individual-focused control condition on type 2 diabetes and CVD biological risk factors (for example, blood pressure and weight) and behavioral risk factors (for example, physical activity and tobacco use). Outcomes are measured at baseline, immediately post-intervention, and at the end of the 12 month period of the study for both groups.

ELIGIBILITY:
Inclusion Criteria:

Primary participants are rural-dwelling Hispanic and non-Hispanic adults who are at-risk for type 2 diabetes or cardiovascular disease and have a family member who is willing to participate if the primary participant is randomly selected to participate with a family member.

Inclusion criteria for the primary participant:

* Is Hispanic or non-Hispanic adult
* Is 18 years of age and older
* Is a primary Spanish or English speaker
* Has internet access
* Has two or more risk factors for type 2 diabetes or cardiovascular disease including:

  1. clinical diagnosis of hypertension;
  2. clinical diagnosis of hyperlipidemia;
  3. clinical diagnosis of prediabetes;
  4. overweight or obese (body mass index ≥ 25 kg/m2);
  5. is a current cigarette smoker;
  6. male 45 years of age or older or female 55 years of age or older;
  7. family history in first degree relative of type 2 diabetes or cardiovascular disease; or
  8. is a female with a history of gestational diabetes mellitus or polycystic ovary syndrome.
* Lives in rural Kentucky
* Is willing to participate in the study for the next 12 months

Inclusion criteria for the co-participating family member if primary participant is randomly selected to participate with a family member

* Is 18 years of age and older
* Is a primary Spanish or English speaker
* Lives in the same household or in close proximity (no further than 25 miles distance) to the primary participant
* Has internet access
* Is willing to participate in the study for the next 12 months

Exclusion Criteria:

Exclusion criteria for family dyads:

Primary participant and family member participant will be excluded if they:

* Have cognitive impairment that preclude them from understanding the consent process, answering questionnaires, or participating in the intervention;
* Have a major psychiatric (e.g., schizophrenia) condition;
* Are pregnant or nursing or plan on becoming pregnant within the next year since dietary needs will be different.

Exclusion criteria that apply only to the primary participant:

* Have known coronary artery or cerebrovascular disease;
* Have a diagnosis of type 1 or type 2 diabetes;
* Have medical contraindications to participate in a lifestyle intervention that includes unsupervised physical activity and weight loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2021-09-11 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-11 (Estimated)

PRIMARY OUTCOMES:
Change in body mass index (BMI) | 1 year (baseline, 3 months and 12 months)
  BMI based on measurements of weight and height and calculated as kg/m2.
Change in blood pressure | 1 year (baseline, 3 months and 12 months)
  Blood pressure assessed using calibrated sphygmomanometry.
Change in lipid profile | 1 year (at baseline, 3 months and 12 months)
  Lipid profile includes LDL-cholesterol, HDL-cholesterol and triglycerides measured using point-of-care testing obtained by fingerstick.
Change in hemoglobin A1c (HbA1c) | 1 year (at baseline, 3 months and 12 months)
  HbA1c will be measured using point-of-care testing obtained by fingerstick.
Change in physical activity level | 1 year (at baseline, 3 months and 12 months)
  Physical activity will be measured using the International Physical Activity Questionnaire (IPAQ) to assess the number of days in the last 7 days that the participant engaged in vigorous or moderate physical activity and confirmed by comparing responses to activity levels as determine through actigraphy.
Change in dietary intake patterns | 1 year (at baseline, 3 months and 12 months)
  Dietary intake patterns will be assessed using the Vioscreen food frequency questionnaire.
Change in tobacco use | 1 year (at baseline, 3 months and 12 months)
  Tobacco use will be confirmed by collection of a saliva sample to determine cotinine levels.

CONTACTS AND LOCATIONS:
Overall Officials: Gia Mudd, RN, PhD, Principal Investigator — University of Kentucky
Locations (1):
- 2201 Regency Rd., Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No